CLINICAL TRIAL: NCT01077557
Title: Fractures Over Time Stratified by HIV Infection and Antiretroviral Therapy (ART) Exposure
Brief Title: Fractures Stratified by HIV and Antiretroviral Therapy (ART) Status
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111950
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Fracture; Infection, Human Immunodeficiency Virus
Keywords: Combivir (Zidovudine+Lamivudine); Trizivir (Abacavir+Lamivudine+Zidovudine); Zidovudine; Epzicom (Abacavir+Lamivudine); Fracture; Amprenavir; human immunodeficiency virus (HIV) infection; antiretroviral (ARV) therapy; Lamivudine; incidence; Abacavir; risk; Fosamprenavir
MeSH Terms: conditions — Fractures, Bone; Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No HIV infection: Subjects without HIV infection (Group 1) are adults, 18 years of age and older, continuously enrolled for at least 12 months in the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database, a health insurance claims database, during the interval between January 1, 1997 and March 31, 2008, and with continuous eligibility for pharmacy benefits. A 3:1 match of subjects without HIV infection to a subject with HIV infection will occur. Each member of the comparator group without HIV infection will be matched on gender, month/year of IHCIS enrolment, and duration of enrollment to the respective study subject with HIV infection.
  Interventions: Other: No Antiretroviral (ARV) Drug Exposure
- HIV infection with no antiretroviral (ARV) drug exposure: HIV infection with no ARV drug exposure (Group 2) represents adults, 18 years of age and older, continuously enrolled for at least 12 months in the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database, a health insurance claims database, during the interval between January 1, 1997 and March 31, 2008, and with continuous eligibility for pharmacy benefits. HIV exposure will be identified by ICD-9-CM code 042 or v08 in one or more diagnostic fields. This group will have no pharmacy dispensing for ARV drugs.
  Interventions: Other: No Antiretroviral (ARV) Drug Exposure
- HIV infection with ARV drug exposure: HIV infection with ARV drug exposure (Group 3) represents adults, 18 years of age and older, continuously enrolled for at least 12 months in the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database, a health insurance claims database, during the interval between January 1, 1997 and March 31, 2008, and with continuous eligibility for pharmacy benefits. HIV exposure will be identified by ICD-9-CM code 042 or v08 in one or more diagnostic fields. This group will have at least one pharmacy dispensing for an HIV antiretroviral drug.
  Interventions: Drug: Any Antiretroviral (ARV) Drug Exposure

INTERVENTIONS:
Other: No Antiretroviral (ARV) Drug Exposure — No pharmacy dispensing of an ARV drug
  Groups: HIV infection with no antiretroviral (ARV) drug exposure; No HIV infection
Drug: Any Antiretroviral (ARV) Drug Exposure — Pharmacy dispensing claim for any ARV drug
  Groups: HIV infection with ARV drug exposure

SUMMARY:
This US population-based study will explore the incidence of and risks for fracture among adults with and without human immunodeficiency virus (HIV) infection. The objectives are to determine the incidence of fracture among persons with and without HIV infection, compare risk factors for fracture among persons with and without HIV infection, and to examine the associations of antiretroviral (ARV) treatment exposure for incidence and risk of fracture among persons with HIV infection.

DETAILED DESCRIPTION:
This study uses data from the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database, a health insurance claims database. The study has two analytic components. The first is a retrospective cohort study comparing subjects without HIV infection to subjects with HIV infection for the incidence of and risk for fracture, including the use of anyARV drugs in persons with HIV infection. The second is a nested case-control study limited to persons with HIV infectiion within the cohort. Cases are those with incident fractures occurring after the diagnosis of HIV infection, and controls those without a fracture. Cases and controls will be compared for risk factors for incident fracture including ARV drug exposure. The drug exposures will include individual nucleoside reverse transcriptase inhibitors (NRTIs) (as permitted by sample size) and the other ARV drug classes.

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria was continuous enrollment for at least 12 months in the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database during the interval between January 1, 1997 and March 31, 2008, age 18 years of age and older, and continuous eligibility for pharmacy benefits during IHCIS enrollment.

Exclusion Criteria:

* Exclusion criteria were membership in the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database without a valid gender or age record, less than 12 months continuous enrolment, and member residence in the 'national' census region. This latter grouping represented members who were either not living in the continental US or were masked for confidentiality reasons based on IHCIS archiving of data per the Health Insurance Portability and Accountability Act.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults (>18 years of age) with and without HIV infection continuously enrolled for at least 12 months in the Integrated Health Care Information Services (IHCIS) National Managed Care Benchmarked Database, a health insurance claims database, during the interval between January 1, 1997 and March 31, 2008, and with continuous eligibility for pharmacy benefits. Health plan enrollees in this database are located in the continental US
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2006-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incident fracture defined by first ICD-9-CM code 733.1 or 800-829 during the follow-up period. Inclusion is restricted to four-digit codes for closed fracture. Exclusions will be codes for skull, face, chest, rib, open fracture, and crushing injuries | From enrollment in IHCIS National Managed Care Benchmarked Database to whichever of the following three event dates comes first: date of first fracture, end date of IHCIS enrollment, or March 31, 2008

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare